CLINICAL TRIAL: NCT01902901
Title: Clinical Implementation of Carrier Status Using Next Generation Sequencing
Acronym: NextGen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 1UM1HG007292-01 (NIH); 1UM1HG007292-01 (NIH)
Record Dates: First submitted 2013-07-10; First posted 2013-07-18 (Estimated); Results first posted 2019-03-13 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Genetic Disorders
Keywords: Whole Genome Sequencing; Carrier status; Genetics
MeSH Terms: conditions — Genetic Diseases, Inborn | interventions — Whole Genome Sequencing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (Active Comparator): Requested carrier status testing.
  Interventions: Genetic: Carrier status testing
- Whole Genome Sequencing (Experimental): These participants will receive the carrier status testing they requested from their provider, plus whole genome sequencing.
  Interventions: Genetic: Whole Genome Sequencing; Genetic: Carrier status testing

INTERVENTIONS:
Genetic: Whole Genome Sequencing — Participants will receive Whole Genome Sequencing
  Arms: Whole Genome Sequencing
Genetic: Carrier status testing — Carrier status testing

SUMMARY:
This study is conducting a randomized controlled trial (RCT) with up to 400 subjects (women & partners) seeking pre-conception carrier testing to assess the impact of the program using Whole Genome Sequencing (WGS).

1. The investigators hypothesize that whole genome sequencing will increase the detection of carrier status for Mendelian recessive and x-linked conditions.
2. The investigators hypothesize that parents will act on the knowledge of their carrier status by making different reproductive choices than parents who do not receive this information.
3. The investigators hypothesize that the psychosocial risks are increased among parents who receive expanded carrier screening using Next Generation Sequencing (NGS) compared with usual care.

DETAILED DESCRIPTION:
Project 1-Clinical Intervention and Outcomes Aim 1: To conduct a randomized controlled trial (RCT) with up to 400 subjects (women & partners) seeking pre-conception carrier testing to assess the impact of the program using Whole Genome Sequencing (WGS).

Aim 2: To develop processes for delivering information from WGS directly into the patient's electronic medical record, and establish innovative reporting strategies that are informative for clinicians and couples acting on this information.

Aim 3: To measure for the integration of sequence information in clinical care for both carrier status and secondary findings including:

1. Patient reported outcomes (PRO) on the impact on quality of life, satisfaction with care, timeliness of reporting, and use of the genomic information.
2. Process outcomes such as timeliness, number of reportable findings, and time of interpretation.

Project 2 -WGS technology, informatics, and Return of Results Committee (RORC)

Aim 1: To generate whole genome sequence and interpret variants on samples randomized from the Kaiser Permanente Northwest (KPNW) preconception carrier screening cohort.

1. To perform whole genome sequencing, assembly, and variant detection for each sample.
2. To provide variant data on each sample with annotation and ranking of clinical significance.
3. To validate data using an orthogonal platform for findings relevant to carrier status and actionable secondary findings.

Aim 2: To develop and implement a return of results committee (RORC) that incorporates evidence to assess criteria for reporting carrier status for reproductive decision making and secondary findings.

Project 3 - Ethical and Psychosocial Implications

Aim 1: To evaluate, patient and clinical perspectives on informational needs, satisfaction, knowledge, and decision-making relating to the choice to obtain results of carrier status from WGS in four categories of genetic conditions.

Aim 2: To evaluate, from patient and clinician perspectives, the immediate and downstream ethical, psychosocial, and behavioral consequences of expanded carrier screening using WGS.

Aim 3: To evaluate the impact of expanded carrier test using WGS on subsequent health care utilization, and to compare the cost of delivery WGS to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Seeking pre-conception carrier status testing or had carrier testing during pregnancy
* Women with a male partner that can be contacted
* Kaiser Permanente Northwest members
* English speaking
* Not currently pregnant

Exclusion Criteria:

* Currently pregnant
* No known or accessible male partner
* Not an English speaker
* Not a Kaiser Permanente member

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 384 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katrina Goddard, PhD, Principal Investigator — Kaiser Permanente; Benjamin Wilfond, MD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Kaiser Permanente Northwest, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Genome sequencing data is shared with dbGaP, and variants are shared with Clinvar.
Time Frame: Ongoing
Access Criteria: Request to dbGaP

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One person consented, but then immediately declined while doing the baseline survey, so she was never randomized.
Period: Overall Study
Arm/Group | Usual Care | Whole Genome Sequencing
Started | 180 | 203
Completed | 180 | 201
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Population: 381 participants completed the baseline survey and had data for analysis. One person in the usual care arm did not complete the baseline survey, and one person in the whole genome sequencing arm completed the baseline survey and then disenrolled from the study a few months later.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Whole Genome Sequencing | Total
Number analyzed (Participants) | 179 | 202 | 381
Age, Categorical [Count of Participants; unit: Participants] — Online survey conducted at the consent visit
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 179 | 202 | 381
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (4.2) | 33 (4.6) | 32 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 179 | 131 | 310
  Male | 0 | 71 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 13 | 25
  Not Hispanic or Latino | 166 | 188 | 354
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 5 | 10 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 2 | 4
  White | 143 | 163 | 306
  More than one race | 26 | 21 | 47
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 159 | 153 | 312

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients That Receive Carrier Testing and Have Results to Return
Description: The investigators will record the number of patients that have both single carrier status testing (usual care) and WGS testing and track how many patients have results to return.
Time Frame: Assessed annually for 4 years, data at the end of the study reported.
Population: All consented participants, including male partners.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Whole Genome Sequencing
Number analyzed (Participants) | 180 | 202
Participants | 9 | 155

2. Secondary Outcome: Patient Satisfaction
Description: Through surveys, interviews, and observations with patients, the investigators will assess their satisfaction with the testing and return of results process.
Time Frame: Assessed annually for 4 years, data at the end of Year 3 reported.
Population: Participants in the usual care arm don't complete satisfaction surveys. Results are WGS arm participants who received genetic testing carrier results in person and reported understanding the information
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Whole Genome Sequencing
Number analyzed (Participants) | 0 | 142
Participants | 0 | 141

3. Other Pre Specified Outcome: Healthcare Utilization
Description: The investigators will evaluate if expanded carrier testing using WGS causes an increase in subsequent health care utilization compared to usual care (typically just cystic fibrosis carrier testing).
Time Frame: The end of Year 4
Population: This data was reported at the end of year 4 for all participants that had at least 6 months of follow-up data.
Measure: Mean (Standard Deviation); unit: Face to face medical encounters
Arm/Group | Usual Care | Whole Genome Sequencing
Number analyzed (Participants) | 177 | 127
Face to face medical encounters | 10 (10) | 10 (9)

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Usual Care | Whole Genome Sequencing
All-Cause Mortality (participants affected / at risk) | 0/180 | 0/203
Serious Adverse Events (participants affected / at risk) | 0/180 | 0/203
Other Adverse Events (participants affected / at risk) | 0/180 | 0/203

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No